CLINICAL TRIAL: NCT00867334
Title: A Phase I/II Study of Gleevec® Combined With Panitumumab (Vectibix®) in Patients Prescreened for C-kit/PDGFr Activated Pathways Using a Proteomic Based Assay
Brief Title: New Individualized Therapy Trial for Metastatic Colorectal Cancer
Acronym: NITMEC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BUS278T
Record Dates: First submitted 2009-03-19; First posted 2009-03-23 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2016-06

CONDITIONS: Colorectal Neoplasm; Colorectal Cancer
Keywords: colorectal neoplasm; colorectal cancer; imatinib mesylate; Gleevec; Physiological Effects of Drugs; panitumumab; Vectibix; c-kit receptor; Receptor; Platelet-Derived Growth Factor alpha
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Imatinib Mesylate; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imatinib mesylate and panitumumab (Experimental): Subjects whose initial liver biopsy samples meet certain lab values will be placed in Arm 1. Each participant assigned to Arm 1 will receive imatinib mesylate for 28 days, followed by a combination of imatinib mesylate and panitumumab.
  Interventions: Drug: Imatinib mesylate and panitumumab
- Panitumumab (standard-of-care) (Active Comparator): Subjects whose initial liver biopsy samples meet certain lab values will be placed in Arm 2. Participants in Arm 2 will receive standard-of-care treatment with panitumumab.
  Interventions: Drug: Standard-of-care treatment with panitumumab

INTERVENTIONS:
Drug: Imatinib mesylate and panitumumab — Patients will be entered into sequential cohorts with escalating doses of imatinib mesylate. After approximately 28 days of monotherapy treatment with imatinib mesylate, patients will be asked to have a liver biopsy performed (this biopsy is voluntary and is not required for continued participation in the study). All patients in this group will then receive imatinib mesylate in combination with standard-of-care doses of panitumumab. After approximately 1-2 months of combination treatment, patients will asked to have an additional liver biopsy performed (this biopsy is voluntary and is not required for continued participation in the study). Combination treatment will continue for the remainder of the subject's time in the trial.
  Other Names: Gleevec; ST1571
  Arms: Imatinib mesylate and panitumumab
Drug: Standard-of-care treatment with panitumumab — Panitumumab as standard of care. After approximately 2-3 months of standard of care treatment, patients will asked to have a liver biopsy performed (this biopsy is voluntary and is not required for continued participation in the study).
  Other Names: Vectibix; ABX-EGF monoclonal antibody
  Arms: Panitumumab (standard-of-care)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of imatinib mesylate in combination with panitumumab for the treatment of stage IV colorectal cancer that has spread to the liver. It will also assess the whether imatinib mesylate, either alone or in combination with panitumumab, is effective in treating this type of cancer. In addition, the study will evaluate the feasibility of a predefined lab score and whether it can predict which patients will respond to treatment with imatinib mesylate.

DETAILED DESCRIPTION:
Recently, a series of clinical trial outcome reports have shown that KRAS mutations (and to a lesser extent KRAS mutations with BRAF V600E mutation) significantly negatively correlate with response to anti-epidermal growth factor (EGFR) mAbs, such as panitumumab, in metastatic colorectal cancer (mCRC) patients. WT KRAS status was shown to be required but not sufficient to confer sensitivity to panitumumab monotherapy. The molecular mechanisms underlying the response or lack of response to EGFR-directed therapies in CRC patients with WT RAS status are unknown. Potential mechanisms of response include activation of EGFR through receptor mutation or autocrine/paracrine ligand binding, activation while tumors that do not respond to EGFR-directed therapy may have activation of other distinct pathways such as VEGF, PDGF, and insulin-like growth factor 1 receptor; activating mutations of additional signaling proteins downstream of EGFR such as PI3K, and Src, or downstream of KRAS, such as RAF; and loss of function genes such as phosphatase and tensin homolog (PTEN). Identifying prognostic and predictive biomarkers to EGFR-directed therapy will prove important for the selection of therapeutic combinations to maximize clinical benefit. In addition to ascertaining resistance mechanisms other biomarkers such as EGFR gene copy number and expression levels of EGFR ligands in tumor cells may be useful to further refine responder population. The current approach applies to the panitumumab monotherapy and indicates that KRAS status should be considered when selecting mCRC patients as candidates for treatment. Thus, patients who are found to harbor KRAS mutation(s) as identified in the pre-treatment liver biopsy specimen will not be eligible for continuation on the trial, but following patient consent, the pre-treatment biopsy will be studied for pathway activation analysis by a CAP/CLIA compliant independent laboratory for research purposes only in the hopes for generating future hypothesis on pathway activation correlating with KRAS mutation status and help extend research into predictive pathway biomarkers for anti-EGFR therapy.

This is a two arm prospective non-randomized study that is designed to assess the safety and efficacy of Gleevec and Vectibix in the treatment of metastatic colorectal cancer to the liver. It also studies the change in phosphorylation levels of Gleevec® targets (PGDT) and tumor burden in patients treated with Gleevec® monotherapy followed by Gleevec® + Vectibix® combination therapy versus treatment with standard of care (panitumumab).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age.
* Histologically documented diagnosis of Stage IV Metastatic Colorectal Cancer with Liver Metastases, refractory or progressive after at least one (1) prior line of therapy that must include a fluoropyrimidine (5-fluorouracil or capecitabine) AND (oxaliplatin OR irinotecan), i.e. FOLFOX, FOLFIRI, XELOX, or XELIRI.
* Documentation of wild type k-Ras expression in the liver lesion.
* At least one measurable site of disease (as defined by Response Evaluation Criteria in Solid Tumors, see Appendix 3), or other response assessment criteria, as appropriate.
* Must have ≥ 1 measurable liver lesion that can be accessed by CT guided biopsy.
* Performance status 0,1, or 2 (ECOG).
* Adequate end organ function, defined as the following: total bilirubin < 1.5 x ULN, SGOT and SGPT < 2.5 x UNL, creatinine < 1.5 x ULN, ANC > 1.5 x 10^9/L, platelets > 100 x 10^9/L.
* Life expectancy of at least 3 months.
* Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 7 days following discontinuation of study drug.
* Written, voluntary informed consent.

Exclusion Criteria:

* Patient has received any other investigational agents within 28 days of first day of study drug dosing, unless the disease is rapidly progressing.
* Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is neither currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
* Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
* Female patients who are pregnant or breast-feeding.
* Patient has a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
* Patient has a known brain metastasis not treated with definitive therapy with stable disease ≥ 4 weeks.
* Patient has known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
* Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
* Patient received chemotherapy within 2 weeks (6 weeks for nitrosourea or mitomycin-C)prior to study entry, unless the disease is rapidly progressing.
* Patient previously received radiotherapy to ≥ 25% of the bone marrow
* Patient had a major surgery within 2 weeks prior to study entry.
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
* Patients intolerant to imatinib mesylate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Edmiston, MD, FACS, Principal Investigator — Inova Fairfax Hospital Cancer Center
Locations (2):
- United States (2):
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Inova Fairfax Hospital Department of Surgery, Falls Church, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at community hospital.
Pre-assignment Details: Inclusion and exclusion criteria for the study were rigid, with only 10 patients of 39 screens being able to enroll. Of these 10 patients, 3 were subsequent withdraws occurring after enrollment of various reasons, thus did not wish to continue to participate in the study.
Groups:
- Treatment With Increasing Doses of Imatinib: Subjects whose initial liver biopsy samples meet certain lab values will be placed in Arm 1. Each participant assigned to Arm 1 will receive imatinib mesylate for 28 days, followed by a combination of imatinib mesylate and panitumumab.
  All patients in this group then received imatinib mesylate in combination with standard-of-care doses of panitumumab.
- Standard of Care Therapy With Panitumumab: Patients entering the control arm (Arm 2) received standard of care therapy with panitumumab (6mg/kg every 2 weeks) until tumor progression. Follow up imaging and biopsy were collected 2-3 months from the beginning of treatment.
Period: Overall Study
Arm/Group | Treatment With Increasing Doses of Imatinib | Standard of Care Therapy With Panitumumab
Started | 6 | 1
Completed | 4 | 0
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment With Increasing Doses of Imatinib | Standard of Care Therapy With Panitumumab | Total
Number analyzed (Participants) | 6 | 1 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (7.9) | 72 (0) | 60.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events
Description: Information about all adverse events, whether volunteered by the subject, discovered by investigator questioning, or detected through physical examination, laboratory test or other means, will be collected and recorded.
Time Frame: From consent up until 4 weeks after patient has stopped study participation
Population: The subject randomized to the "Standard of Care Therapy with Panitumumab arm" withdrew after randomization, so no data was collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Increasing Doses of Imatinib | Standard of Care Therapy With Panitumumab
Number analyzed (Participants) | 6 | 0
Participants | 5 | 0

2. Secondary Outcome: Number of Participants With Stabilization or Reduction in Tumor Size
Description: Results reported as number of patients with stabilization or reduction in tumor size. Tumor response is defined by the Response Evaluation Criteria in Solid Tumors (RECIST) solid tumor response criteria, evaluated by CT.
Time Frame: 8 weeks after baseline
Population: CT measurements of metastasis were planned through timepoint 3 (24 weeks). One participant only had data at timepoint 1 (8 weeks), so timepoint 1 was chosen as the post-treatment comparison timepoint for all participants. One subject in the imatinib group and one subject in the panitumumab group withdrew before obtaining 8 week evaluations.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Increasing Doses of Imatinib | Standard of Care Therapy With Panitumumab
Number analyzed (Participants) | 5 | 0
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: Any serious adverse event occurring after the patient has provided informed consent, has started taking the study medication, and until 4 weeks after the patient has stopped study participation.
Description: Note that the subject randomized to the standard of care arm withdrew after randomization, so adverse event data is not available.
Arm/Group | Treatment With Increasing Doses of Imatinib | Standard of Care Therapy With Panitumumab
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/0
Other Adverse Events (participants affected / at risk) | 5/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Increasing Doses of Imatinib (N=6) | Standard of Care Therapy With Panitumumab (N=0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Hemorrhage/Bleeding (General disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Increasing Doses of Imatinib (N=6) | Standard of Care Therapy With Panitumumab (N=0)
Rash or injection site reaction (Skin and subcutaneous tissue disorders) | 3 (12) | 0 (0)
Priuritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hemorrhage GU - Vaginal (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Edema (Blood and lymphatic system disorders) | 4 (9) | 0 (0)
Infection (Renal and urinary disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 2 (5) | 0 (0)
Weakness (General disorders) | 1 (1) | 0 (0)
Generalized aches and pain (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dehydration (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Creatinine (General disorders) | 1 (8) | 0 (0)
Alkaline Phosphatase (General disorders) | 3 (21) | 0 (0)
Alanine aminotransferease (General disorders) | 3 (8) | 0 (0)
Hemoglobin (General disorders) | 3 (11) | 0 (0)
Fever (General disorders) | 1 (2) | 0 (0)
Liver dysfunction (Hepatobiliary disorders) | 1 (2) | 0 (0)
Total Bilirubin (General disorders) | 1 (3) | 0 (0)
Aspartate aminotransferase (General disorders) | 2 (6) | 0 (0)
Mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypokalemia (General disorders) | 1 (1) | 0 (0)
Proteinuria (General disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Rigors/chills (General disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Absolute neutrophil count (General disorders) | 1 (1) | 0 (0)
Platelets (General disorders) | 1 (2) | 0 (0)
Glucose (General disorders) | 1 (2) | 0 (0)
Anal Incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Stool in urine (Renal and urinary disorders) | 1 (3) | 0 (0)
Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fistula - bladder and rectum (Renal and urinary disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Albumin (General disorders) | 1 (8) | 0 (0)
White Blood Count (Blood and lymphatic system disorders) | 1 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
This is a pilot study utilizing only a small sample size of people.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No